CLINICAL TRIAL: NCT06777264
Title: Clinical Study on Inaticabtagene Autoleucel (Inati-cel; CNCT19) Injection for Adolescents and Adults With B-Cell Acute Lymphoblastic Leukemia in First Complete Remission (CR1)
Brief Title: Inaticabtagene Autoleucel (Inati-cel; CNCT19) Treatment for Newly Diagnosed B-cell ALL Patients in CR1
Acronym: JUVENTAS-ALL05
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2024]TXB ethic review NO.023
Record Dates: First submitted 2024-12-31; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Acute Lymphoblastic Leukemia; B Cell ALL
Keywords: Chimeric Antigen Receptor T (CAR-T)Cell; Acute Lymphoblastic Leukemia; B-ALL; Inaticabtagene Autoleucel
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Biological Products

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological: Inaticabtagene autoleucel (Experimental): Administration of Inaticabtagene Autoleucel (CD19 CAR-T cells) in newly diagnosed B-ALL patients aged 14 to 70 years in their first complete remission (CR1).
  Interventions: Biological: Biological: single dose of Inaticabtagene autoleucel

INTERVENTIONS:
Biological: Biological: single dose of Inaticabtagene autoleucel — Inaticabtagene autoleucel will be transfusioned intravenously at the recommended dose of 0.5×10^8 (ranging 0.2-0.6×10^8) viable CAR-T cells.
  Other Names: Inati-cel; CNCT-19

SUMMARY:
This investigator-initiated, prospective, single-arm, open-label, single-center phase II study aims to evaluate the long-term survival benefit and safety of a commercial CD19 CAR-T product in newly diagnosed Philadelphia chromosome-positive or negative (Ph-positive or Ph-negative) B-cell ALL patients who achieve CR1 after induction chemotherapy. A total of 20 patients will be enrolled in the study. The primary endpoints include disease-free survival (DFS) and overall survival (OS) rates after a median follow-up of 2 years, minimal residual disease (MRD) negativity rate, and the proportion of patients undergoing subsequent hematopoietic stem cell transplantation (HSCT). The frequency and severity of adverse events (AEs) and serious adverse events (SAEs) occurring after infusion will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥14 years and ≤70 years at screening, with no restrictions on gender.
2. ECOG performance status of 0 to 1.
3. Newly diagnosed B-ALL within 12 months and achieving CR1 after standard induction chemotherapy. This includes B-ALL patients with <5% bone marrow blasts, no blasts in peripheral blood, and no extramedullary leukemia. Diagnosis and chemotherapy regimen follow the Chinese Guidelines for Diagnosis and Treatment of Adult Acute Lymphoblastic Leukemia (2021 Edition).
4. At the time of B-ALL diagnosis, leukemia cells in bone marrow or peripheral blood confirmed as CD19-positive via flow cytometry.
5. Adequate organ function meeting the following criteria:

   1. Aspartate aminotransferase (AST) ≤3× upper limit of normal (ULN).
   2. Alanine aminotransferase (ALT) ≤3× ULN.
   3. Total bilirubin ≤2× ULN (for patients with Gilbert's syndrome, total bilirubin ≤3.0× ULN and direct bilirubin ≤1.5× ULN).
   4. Serum creatinine ≤1.5× ULN, or creatinine clearance ≥60 mL/min (calculated using the Cockcroft-Gault formula).
   5. International Normalized Ratio (INR) ≤1.5× ULN and activated partial thromboplastin time (APTT) ≤1.5× ULN.
   6. Minimum pulmonary reserve defined as ≤Grade 1 dyspnea and oxygen saturation >91% on room air.
6. No intent or eligibility for hematopoietic stem cell transplantation.
7. Meets the leukapheresis standards of the study center, with no contraindications for apheresis.
8. Women of childbearing potential must have a negative blood/urine pregnancy test during the Inati-cel screening period and before preconditioning (results within three days prior to preconditioning). All male and female patients of childbearing potential must agree to use effective contraception throughout the study and for at least two years following study treatment. A female is considered of childbearing potential if biologically capable of having children and engaging in regular sexual activity. Women are considered not of childbearing potential if they meet at least one of the following:

   1. History of hysterectomy, bilateral oophorectomy, or bilateral tubal ligation.
   2. Medically confirmed ovarian failure.
   3. Postmenopausal (absence of menstruation for at least 12 consecutive months).

Exclusion Criteria:

1. Diagnosis of Burkitt lymphoma/leukemia, heterozygous or double-hit leukemia, or chronic myeloid leukemia in blast crisis.
2. Presence of ≥5% blasts in the bone marrow or peripheral blood, or evidence of extramedullary leukemia before screening or preconditioning.
3. Prior treatment with CAR-T cell therapy or hematopoietic stem cell transplantation (HSCT) before screening or preconditioning.
4. Genetic syndromes associated with bone marrow failure, including Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or other known bone marrow failure syndromes.
5. Presence of any of the following conditions:

   1. Positive for HBsAg and/or HBeAg.
   2. Positive for HBe-Ab and/or HBc-Ab with HBV-DNA levels above the detectable threshold.
   3. Positive for HCV-Ab.
   4. Positive for TP-Ab.
   5. EBV-DNA or CMV-DNA levels above the detectable threshold.
   6. Positive for HIV antibodies.
6. Diagnosis of other malignancies within the past 5 years, unless the tumor was curatively treated, with a follow-up period exceeding 5 years, and a low risk of recurrence as assessed by the investigator.
7. Presence of any of the following cardiac conditions:

   1. Left ventricular ejection fraction (LVEF) ≤45%.
   2. Congestive heart failure classified as NYHA class III or IV.
   3. Severe arrhythmias requiring treatment or clinically significant conduction abnormalities on ECG, including QTc ≥480 ms (QTcB = QT/RR^1/2).
   4. Uncontrolled hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg) or pulmonary hypertension despite standard treatment.
   5. Unstable angina.
   6. Myocardial infarction or coronary artery bypass/stent surgery within the past 6 months.
   7. Clinically significant valvular disease.
   8. Other cardiac conditions deemed unsuitable for study enrollment by the investigator.
8. History of epilepsy, ischemic or hemorrhagic stroke, cerebellar disease, or other active central nervous system disorders.
9. Clinically significant pleural effusion at the time of screening.
10. History of deep vein thrombosis or pulmonary embolism within the past 6 months.
11. Known hypersensitivity to any components of the investigational products used in the trial.
12. Receipt of live vaccines within 6 weeks prior to screening.
13. Presence of active infections at the time of screening.
14. An expected survival of less than 3 months.
15. Participation in other interventional clinical studies involving investigational drugs:

    1. For investigational drugs not yet approved, the last dose administered less than 3 months before cell infusion.
    2. For approved drugs, the last dose administered less than 5 half-lives before cell infusion.
16. Any other conditions deemed unsuitable for study participation by the investigator.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
2-year DFS rate (2yDFSR) | Up to 2 years
  The proportion of patients who remain free from bone marrow disease relapse or death from any cause, assessed after a median follow-up of 2 years
2-year OS rate (2yDFSR) | Up to 2 years
  The proportion of patients who remain alive after a median follow-up of 2 years
DFS | Up to 2 years
  The time from Inati-cel infusion to morphological relapse of B-ALL in the bone marrow, or death from any cause (whichever occurs first).
OS | Till the end of the study, up to 5 years
  The time from Inati-cel infusion to death from any cause

SECONDARY OUTCOMES:
Proportion of patient underwent subsequent hematopoieticstem cell transplantation | Till the end of the study, up to 5 years
  Proportion of patient underwent subsequent hematopoieticstem cell transplantation
MRD negativity rate | 6 months
  the proportion of patients achieved undetectable levels of minimal residual disease at Day 28、Month 2，3，6 by flow cytometry and at Day 28 by NGS
Maximum observed concentration(Cmax) | 6 months
Time of Cmax (Tmax) | 6 months
Partial area under the concentration-time curve (from time zero to 28days after dosing , AUC 0-28 day) | 6 months

IPD SHARING:
Plan to Share IPD: Undecided